CLINICAL TRIAL: NCT00036920
Title: Phase II Study Of TLK286 For The Treatment Of Advanced Non-Small Cell Lung Cancer
Brief Title: TLK286 in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TLK-286.2004; MSKCC-01147; CDR0000069341 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2063
Record Dates: First submitted 2002-05-13; First posted 2003-11-21 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — TER 286

INTERVENTIONS:
Drug: canfosfamide hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of TLK286 in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the 12-month survival of patients with advanced non-small cell lung cancer treated with TLK286. II. Determine the overall survival of patients treated with this drug. III. Determine the objective response rate, duration of objective response, time to tumor progression, and disease stabilization in patients treated with this drug. IV. Determine the safety of this drug in these patients.

OUTLINE: This is a multicenter study. Patients receive TLK286 IV over 30 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks for 1 year and then every 12 weeks thereafter.

PROJECTED ACCRUAL: Approximately 55 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed non-small cell lung cancer (NSCLC), including: Squamous cell carcinoma Undifferentiated carcinoma Adenocarcinoma Mixed (i.e., adenocarcinoma with squamous cell carcinoma) No mixed tumors containing small cell lung carcinoma elements Bronchoalveolar carcinoma Large cell carcinoma Bronchoalveolar lavage allowed for diagnosis Advanced or metastatic NSCLC Stage IIIB disease ineligible for combined chemotherapy and radiotherapy OR Stage IV disease Progressive NSCLC during or after first-line therapies with platinum-containing chemotherapy regimens in the advanced or metastatic setting Measurable disease by radiological imaging techniques Previously treated CNS metastases allowed provided: Neurologically stable Oral or IV steroids or anticonvulsants not required No active disease by CT scan or MRI No known leptomeningeal metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.0 mg/dL ALT and AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min No gross hematuria Cardiovascular: No uncontrolled cardiac arrhythmia No myocardial infarction within the past 6 months Other: No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer No severe concurrent disease, infection, or comorbidity that would preclude study No other unstable medical conditions No psychiatric disorders that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy At least 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF) No concurrent immunotherapy No concurrent biological response modifiers Chemotherapy: See Disease Characteristics No more than 2 prior cytotoxic regimens in the advanced or metastatic setting At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas and mitomycin) No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy At least 4 weeks since prior radiopharmaceuticals At least 2 weeks since prior palliative radiotherapy No concurrent radiotherapy except local radiotherapy for pain or solitary brain metastasis if not progressing systemically Surgery: At least 4 weeks since prior major surgery Other: Recovered from prior therapy Prior adjuvant therapy allowed At least 30 days since prior investigational drugs No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2002-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark G. Kris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Henner WD, Figlin RA, Garland LL, et al.: Phase 2 study of TLK286 (GST P1-1 activated glutathione analog) in advanced non-small cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1249, 2002.